CLINICAL TRIAL: NCT05481502
Title: A Prospective Trial to Evaluate Immune Determinants of the Response and the Toxicity to Adoptive Cell Therapy (ACT) in Solid and Hematologic Tumors
Brief Title: An Exploratory Study to Evaluate Immune Determinants of the Response to Adoptive Cell Therapy (ACT) in Solid and Hematologic Tumors
Acronym: PIONEER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A00472-41; 2022/3404 (Other: CSET number)
Record Dates: First submitted 2022-06-24; First posted 2022-08-01 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor, Adult; Solid Tumor, Childhood; Hematologic Cancer
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving advanced therapy medicinal products (Experimental)
  Interventions: Procedure: Tumor biopsy; Procedure: Blood sample; Procedure: Bone marrow sample

INTERVENTIONS:
Procedure: Tumor biopsy — 3 biopsies will be collected: at baseline, at day+15 and optionally at relapse
Procedure: Blood sample — 7 blood samples (25ml) will be taken: at day-7 before treatment start, at day0, at day+3, day+7, day+15, month+3 and at relapse
Procedure: Bone marrow sample — If a bone marrow biopsy or aspiration is performed as part of routine care, 1 mL of bone marrow aspiration or one more biopsy will be sampled

SUMMARY:
This is a study to explore the phenotypic and transcriptional changes of different cellular components in the tumor following the injection of somatic cell therapy drugs.

The second objective is to explore phenotypic and transcriptional changes of different cellular components in blood and bone marrow following injection of somatic cell therapy drugs.Then correlate the phenotypic and transcriptional profile of different tumor, blood and bone marrow immune populations with clinical response and/or toxicity. And to finish this study is designed in order to identify a phenotypic, transcriptional and epigenetic profile of intra-tumoral adoptive cells and correlate this profile with clinical response and/or toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated to a social security regimen
* Tumor lesion accessible to core biopsies
* Patient who is fully informed, able to comply with the protocol and who signed the informed consent
* Pediatric patients > than 2 years old can be included
* No restriction about the Eastern Cooperative Oncology Group (ECOG) status

Exclusion Criteria:

* Coagulation abnormality prohibiting a biopsy (but patients can still give their consent for blood and bone marrow samples).
* Tumor lesion not accessible to core biopsies.
* Pregnant or nursing women cannot participate in this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of frequency, phenotype and transcriptional profile of the different immune subsets in the tumor following adoptive cell therapy infusion using spectral flow cytometry and RNA sequencing | 3 months following ACT

SECONDARY OUTCOMES:
Objective Response | 3 months following ACT
  Defined by RECIST 1.1 score for lymphoma and solid tumors
Progression-free survival | 5 years after first ACT infusion
  Defined as the time between the adoptive cell therapy and progression, or death whatever the cause, whichever occurs first.
Overall survival | 5 years after first ACT infusion
  Defined as the time between the adoptive cell therapy injection and death whatever the cause
Safety of biopsies procedures (when applicable) graded according to CTCAE v5.0 | From enrollment to 30 days after the last sample

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val De Marne, France